CLINICAL TRIAL: NCT04699396
Title: The Immediate Effect of Two Mobilization With Movement Techniques on Dorsiflexion, Dynamic Balance and Performance Variables, in Futsal Athletes With Chronic Ankle Instability: A Randomized Controlled Trial
Brief Title: The Immediate Effect of Mobilisation With Movement in Amateur Futsal Athletes With Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Alexandre Portela, Principal Investigator, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESS-MWM
Record Dates: First submitted 2020-12-30; First posted 2021-01-07 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Ankle Injuries and Disorders
MeSH Terms: conditions — Ankle Injuries; Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mobilisation with Movement 1 (MWM1) (Experimental): Participants received two ankle dorsiflexion MWM techniques, with glides applied at fibula and talus. Three sets of 10 repetitions of each techniques, were administrated.
  Interventions: Procedure: Mobilisation With Movement 1
- Mobilisation with Movement 2 (MWM2) (Experimental): Participants received two ankle dorsiflexion MWM techniques, with glides applied at talus and fibula (order of application inverted). Three sets of 10 repetitions of each techniques, were administrated.
  Interventions: Procedure: Mobilisation With Movement 2
- Placebo (Placebo Comparator): The Placebo group participants performed the same number of sets and repetitions of lean/lunge forward into dorsiflexion, without any glide application, in the same position
  Interventions: Other: Placebo
- Intervention (Experimental): The experimental groups (MWM1 and MWM2), were later merged into a single Intervention group.
  Interventions: Procedure: Mobilisation With Movement 1; Procedure: Mobilisation With Movement 2

INTERVENTIONS:
Procedure: Mobilisation With Movement 1 — Application of a sustained passive accessory movement to a joint (talus or fibula) while the patient actively performs a forward lean/lunge that was previously limited.
  3 sets of 10 repetitions of a glide applied to the talus were performed, followed by 3 sets of 10 repetitions of a glide applied to the fibula.
  Other Names: Mulligan
  Arms: Intervention; Mobilisation with Movement 1 (MWM1)
Procedure: Mobilisation With Movement 2 — Application of a sustained passive accessory movement to a joint (talus or fibula) while the patient actively performs a forward lean/lunge that was previously limited.
  3 sets of 10 repetitions of a glide applied to the fibula were performed, followed by 3 sets of 10 repetitions of a glide applied to the talus.
  Other Names: Mulligan
  Arms: Intervention; Mobilisation with Movement 2 (MWM2)
Other: Placebo — The Placebo group participants performed the same number of sets and repetitions (6 sets of 20 repetitions) of lean/lunge forward into dorsiflexion, without any glide application.
  Arms: Placebo

SUMMARY:
Chronic ankle instability (CAI) is an increasingly prevalent condition among futsal athletes. Mobilization with Movement (MWM) is a conservative rehabilitation strategy commonly used in this condition. Even so, the effects of two MWM dorsiflexion techniques on sports performance are not known. The aim is to analyze the immediate effect of two MWM techniques on the dorsiflexion range of motion, the dynamic balance and the performance variables in futsal athletes with CAI. Also, to analyze the impact of performing them in a different order.

ELIGIBILITY:
Inclusion Criteria:

1. A history of at least one significative ankle sprain:

   * Initial sprain must have occurred at least 12 months prior to study enrolment;
   * Was associated with inflammatory symptoms;
   * Created at least one interrupted day of desired physical activity;
   * The most recent injury must have occurred more than 3 months prior to study enrolment.
2. A history of the previously injured ankle joint "giving way" and/or recurrent sprain and/or "feelings of instability":

   * Participants should report at least two episodes of "giving way" in the 12 months prior to study enrolment, to account for the seasonal nature of futsal;
   * Recurrent sprain was defined as two or more sprains to the same ankle.
3. Self-reported ankle instability should be confirmed with the Ankle Instability Instrument: answer "yes" to at least 5 yes/no questions.

Exclusion Criteria:

1. A history of previous surgeries to the musculoskeletal structures (i.e., bones, joint structures, nerves) in either lower extremity.
2. A history of bilateral ankle sprain.
3. A history of a fracture in either lower extremity requiring realignment.
4. Acute injury to musculoskeletal structures of other joints of the lower extremity in the previous 3 months that impacted joint integrity and function (i.e., sprains, fractures), resulting in at least one interrupted day of desired physical activity.
5. Have conditions for which manual therapy is generally contraindicated (such as the presence of a tumour, fracture, rheumatoid arthritis, osteoporosis, prolonged history of steroid use, or severe vascular disease).
6. Receiving concurrent physiotherapy treatment in the last 3 months.
7. Inability to read Portuguese.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Dorsiflexion range of motion | Immediate after procedure
  The dorsiflexion range of motion (DFROM) of the ankle joint was measured by the Weight-Bearing Lunge Test (WBLT)

SECONDARY OUTCOMES:
Dynamic balance | Immediate after procedure
  The dynamic balance was measured by the anterior (ANT), posteromedial (PM) and posterolateral (PL) reach directions of the Star Excursion Balance Test (SEBT)
Performance variables | Immediate after procedure
  The performance variables were measured by the time needed to complete the Side Hop Test and the Sprint Test

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Superior de Saúde do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lopez-Segovia M, Vivo Fernandez I, Herrero Carrasco R, Pareja Blanco F. Preseason Injury Characteristics in Spanish Professional Futsal Players: The LNFS Project. J Strength Cond Res. 2022 Jan 1;36(1):232-237. doi: 10.1519/JSC.0000000000003419. PMID 31895285
- [Background] Hertel J, Corbett RO. An Updated Model of Chronic Ankle Instability. J Athl Train. 2019 Jun;54(6):572-588. doi: 10.4085/1062-6050-344-18. Epub 2019 Jun 4. PMID 31162943
- [Background] Cruz-Diaz D, Lomas Vega R, Osuna-Perez MC, Hita-Contreras F, Martinez-Amat A. Effects of joint mobilization on chronic ankle instability: a randomized controlled trial. Disabil Rehabil. 2015;37(7):601-10. doi: 10.3109/09638288.2014.935877. Epub 2014 Jul 3. PMID 24989067
- [Background] Langarika-Rocafort A, Emparanza JI, Aramendi JF, Castellano J, Calleja-Gonzalez J. Intra-rater reliability and agreement of various methods of measurement to assess dorsiflexion in the Weight Bearing Dorsiflexion Lunge Test (WBLT) among female athletes. Phys Ther Sport. 2017 Jan;23:37-44. doi: 10.1016/j.ptsp.2016.06.010. Epub 2016 Jun 29. PMID 27665249
- [Background] Marron-Gomez D, Rodriguez-Fernandez AL, Martin-Urrialde JA. The effect of two mobilization techniques on dorsiflexion in people with chronic ankle instability. Phys Ther Sport. 2015 Feb;16(1):10-5. doi: 10.1016/j.ptsp.2014.02.001. Epub 2014 Feb 14. PMID 24679362
- [Background] Gribble PA, Delahunt E, Bleakley C, Caulfield B, Docherty CL, Fourchet F, Fong D, Hertel J, Hiller C, Kaminski TW, McKeon PO, Refshauge KM, van der Wees P, Vicenzino B, Wikstrom EA. Selection criteria for patients with chronic ankle instability in controlled research: a position statement of the International Ankle Consortium. J Orthop Sports Phys Ther. 2013 Aug;43(8):585-91. doi: 10.2519/jospt.2013.0303. Epub 2013 Jul 31. PMID 23902805